CLINICAL TRIAL: NCT00533468
Title: "Lidocaine 4% Cream (LMX4) vs Placebo for Pain Due to Lumbar Puncture in Infants 0-60 Days of Age."
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Ferndale Laboratories, Inc. (Industry)
Responsible Party: Principal Investigator, James Reingold, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 05-130
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Pain
Keywords: pain; lumbar puncture; neonates; infants; emergency department; topical anesthesia; LMX4
MeSH Terms: conditions — Pain; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Drug (Experimental): Active 4% Lidocaine topical cream (LMX4 cream) applied under occlusive dressing
  Interventions: Drug: Lidocaine Cream 4%
- Placebo (Placebo Comparator): Placebo Cream made on same run at factory but without active Lidocaine 4% drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Cream 4% — Topical cream, 2g applied under occlusive dressing for 20 minutes prior to the procedure
  Other Names: LMX4
  Arms: Active Drug
Drug: Placebo — inactive placebo without LMX4
  Arms: Placebo

SUMMARY:
The study's hypothesis is LMX4 cream, a topical anesthetic cream, will reduce the pain of infants undergoing Lumbar Puncture (spinal tap).

DETAILED DESCRIPTION:
Pain of infants will be measured using the Neonatal Facial Coding System by videotaping the infant's face while they undergo the procedure. A comparison between the group that received active drug and the group that received placebo will allow a measurement of the difference, if any, of the pain experienced during the procedure of the infants.

ELIGIBILITY:
Inclusion Criteria:

* Full term (>=37 weeks gestation)
* Age 0-60 Days
* Undergoing Lumbar Puncture

Exclusion Criteria:

* Unstable
* Premature (<37 weeks gestation)
* Allergy to study medicine
* Parent refusal of consent

Ages: 0 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Reingold, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- Women's and Children's Hospital of Buffalo, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: patients in this arm were randomized to placebo in a double blind fashion
- Active Drug: patients in this arm were randomized to receive the active drug, LMX4, in a double blind fashion
Period: Overall Study
Arm/Group | Placebo | Active Drug
Started | 35 | 35
Completed | 28 | 24
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Placebo; Active Drug: patients were randomized to placebo or active drug in a double blind fashion
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 24 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 33.6 (16.3) | 28.2 (14.9) | 31.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 17 | 12 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 18 | 6 | 24
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 5 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52
gestational age [Mean (Standard Deviation); unit: weeks] | 39.4 (1.3) | 38.8 (1.2) | 39 (1.2)
WEIGHT [Mean (Standard Deviation); unit: GRAMS] | 5094 (2147) | 4492 (1387) | 4708 (1651)

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Facial Coding System Score
Description: 10 measures of pain, all scored 0 or 1, high score means more pain. No pain would be recorded as zero, maximum pain recorded as 10
Time Frame: Score was measured at baseline, upon positioning for the procedure, immediately prior to needle insertion, during needle insertion, 1 minute post-needle insertion, and post-procedure when the infant had recovered from the procedure and was swaddled
Population: infants 0-60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: patients were randomized to placebo in this arm in a double blind fashion
- Active Drug: patients were randomized active drug in this arm in a double blind fashion
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 28 | 24
score on a scale
  Baseline | 4.6 (4) | 3.9 (3.5)
  Positioning | 8.3 (5) | 8 (4.5)
  Pre-needle | 7.6 (6) | 6.7 (5)
  Needle Insertion | 9.3 (6) | 9.9 (5.5)
  Post-needle Insertion | 5.7 (6.5) | 6.1 (6)
  Post-procedure | 4.2 (8.5) | 5.9 (8)

2. Secondary Outcome: Time of Procedure
Description: Time, measured in minutes, required to complete procedure from infant's presentation to the Emergency Department
Time Frame: Infant's stay in the Emergency Department
Population: infants 0-60 days of age
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Active Drug: patients were randomized to active drug in this arm in a double blind fashion
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 28 | 24
minutes | 31 (12) | 36 (16)

3. Secondary Outcome: Percentage of Procedures With Success
Description: Whether the Lumbar Puncture resulted in recovery of spinal fluid that could be sent for usual testing
Time Frame: During patient's Emergency Department Stay
Measure: Number; unit: percentage of procedures
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 28 | 24
percentage of procedures | 96 | 75

ADVERSE EVENTS:
Groups:
- Placebo: Patients in this arm were administered placebo without active drug
- Active Drug: patients in this arm were administered active drug
Arm/Group | Placebo | Active Drug
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24
Other Adverse Events (participants affected / at risk) | 10/28 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Active Drug (N=24)
rash (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)

LIMITATIONS AND CAVEATS:
Significant technical limitation was encountered regarding videotaping of infant faces when properly positioned for the procedure, as the research assistant had to be underneath the nurse's arm with the camera adjacent to the nurse's breast. This resulted in many exclusions of patients enrolled by the male research assistants as the camera was not in proper position. The many exclusions reduced the study's power to reach a statistically significant difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No